CLINICAL TRIAL: NCT03600779
Title: Application of the Inhomogeneous Magnetisation Transfer MRI (ihMT) Technique, a New Myelin-specific MRI Technique, in Multiple Sclerosis
Brief Title: Application of ihMT MRI in Multiple Sclerosis
Acronym: ihMTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-61
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sclerosis, Multiple
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sequence Analysis, DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental group 1.5T (Experimental): Population of patients with myelin syndrome (MS) at the the disease onset with active lesions inhomogeneous Magnetisation Transfer (ihMT) sequence will be performed.
  Interventions: Device: inhomogeneous Magnetisation Transfer (ihMT) sequence
- control group 1.5 T (Active Comparator): healthy volunteers matched in sex and age inhomogeneous Magnetisation Transfer (ihMT) sequence will be performed.
  Interventions: Device: inhomogeneous Magnetisation Transfer (ihMT) sequence
- experimental group 3T (Experimental): Population of patients with myelin syndrome (MS) at the the disease onset with active lesions inhomogeneous Magnetisation Transfer (ihMT) sequence at 3T will be performed.
  Interventions: Device: inhomogeneous Magnetisation Transfer (ihMT) sequence at 3T
- control group 3T (Active Comparator): inhomogeneous Magnetisation Transfer (ihMT) sequence will be performed. inhomogeneous Magnetisation Transfer (ihMT) sequence at 3T will be performed.
  Interventions: Device: inhomogeneous Magnetisation Transfer (ihMT) sequence at 3T

INTERVENTIONS:
Device: inhomogeneous Magnetisation Transfer (ihMT) sequence — robust technique has shown great sensitivity for evaluating the demyelination processes using MRI at 1.5T
  Arms: control group 1.5 T; experimental group 1.5T
Device: inhomogeneous Magnetisation Transfer (ihMT) sequence at 3T — robust technique has shown great sensitivity for evaluating the demyelination processes using MRI at 3T
  Arms: control group 3T; experimental group 3T

SUMMARY:
The development of in vivo biomarkers sensitive to myelin disruption represents a major clinical need to be able to monitor the demyelination processes as well as the effect of remyelinating therapies in multiple sclerosis. The investigators recently proposed a technique, derived from the conventional magnetisation transfer (MT): inhomogeneous Magnetisation Transfer (ihMT). In preliminary studies, this simple-to-implement and robust technique has shown great sensitivity for evaluating the demyelination processes. The goal of the project is to evaluate the ability of ihMT to measure and describe the spontaneous demyelination and remyelination processes involved in active lesions in a population of patients with MS at the the disease onset.

DETAILED DESCRIPTION:
The development of in vivo biomarkers sensitive to myelin disruption (demyelination and remyelination) represents a major clinical need to be able to monitor the demyelination processes as well as the effect of remyelinating therapies in multiple sclerosis. The investigators recently proposed a technique, derived from the conventional magnetisation transfer (MT): inhomogeneous Magnetisation Transfer (ihMT). In preliminary studies, this simple-to-implement and robust technique has shown great sensitivity for evaluating the demyelination processes. The goal of the project is to evaluate the ability of ihMT to measure and describe the spontaneous demyelination and remyelination processes involved in active lesions in a population of patients with MS at the the disease onset.

ELIGIBILITY:
Inclusion Criteria:

* For Patients and Controls :

  * Adult patient, male and female, age 18 to 45
  * Patient affiliated with health insurance coverage,
  * Patient who signed a free and informed consent after receiving detailed, understandable and honest information,
* For patients only :

  * Patient with relapsing-remitting multiple sclerosis according to the McDonald 2010 criteria
  * Disease duration of less than 5 years
  * Patients treated or not treated with first-line disease modifying therapy
  * Detection of at least one post-Gadolinium injection active lesion identified on the initial brain MRI (T0)

Exclusion Criteria:

* For patients only :

  • Patients with a progressive form of MS other than the early relapsing-remitting form (primary progressive or secondary progressive)
* For Patients and Controls :

  * Patients with the usual contraindications for MRI (pacemaker, agitation, metal shards, claustrophobia)
  * Patients at risk of non-compliance to the exam: basic problems with understanding, confusion, involuntary movements, poor tolerance of prolonged supine position
  * Patients who are unable to give their consent: problems with understanding, lack of vigilance, confusion
  * Woman who is pregnant and breastfeeding
  * Patients with a history of neurological or psychiatric condition
  * Patients under guardianship or trusteeship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
ihMTR ratio at 1.5TMRI | 1 year
  ihMT 3D technique at 1.5TMRI on active lesions with baseline measurements
Magnetic transfert (MT) at 1.5TMRI | 1 year
  relative signal variations of the conventional magnetization transfer (MT)
Myelin water fraction at 1.5TMRI | 1 year
  myelin water fraction (MWF), an MRI biomarker of myelin, in new MS lesions

SECONDARY OUTCOMES:
ihMTR ratio at 3TMRI | 1 year
  Relative variations in ihMTR ratio measured at 3T will be compared to those measured at 1.5T at the same points in time to opmtimize 3D ihMT technique at 3TMRI
Evaluate the predictive value of ihMT | 1 year
  Evaluate the predictive value of the measured dynamics with respect to the final progression of the lesions

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hotipaux de Marseille, Marseille, PACA, France